CLINICAL TRIAL: NCT01641666
Title: An Open-Label Study to Assess the Safety and Tolerability of Boceprevir in Combination With Peginterferon Alfa-2b Plus Ribavirin for Treatment of Vietnamese Subjects With Chronic Hepatitis C Genotype 1 Who Failed Prior Treatment With Any Interferon Plus Ribavirin in Vietnam
Brief Title: Safety and Tolerability of Boceprevir in Combination With Peginterferon Alfa-2b Plus Ribavirin for the Treatment of Vietnamese Subjects With Chronic Hepatitis C Genotype 1 (P08599)
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P08599
Record Dates: First submitted 2012-07-11; First posted 2012-07-17 (Estimated); Last update posted 2015-09-09 (Estimated); Status verified 2015-09

CONDITIONS: Chronic Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — N-(3-amino-1-(cyclobutylmethyl)-2,3-dioxopropyl)-3-(2-((((1,1-dimethylethyl)amino)carbonyl)amino)-3,3-dimethyl-1-oxobutyl)-6,6-dimethyl-3-azabicyclo(3.1.0)hexan-2-carboxamide; peginterferon alfa-2b; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Peg2b + Ribavirin + Boceprevir (Experimental): Peginterferon alpha-2b (Peg2b) plus ribavirin (RBV) starting on Day 1 and boceprevir starting on Week 5
  Interventions: Drug: Boceprevir; Drug: Peginterferon Alfa-2b 1.5 mcg/kg/week; Drug: Ribavirin

INTERVENTIONS:
Drug: Boceprevir — Boceprevir will be dosed orally at a dose of 800 mg three times daily (TID) for a total daily dose of 2400 mg.
  Other Names: SCH 503034
Drug: Peginterferon Alfa-2b 1.5 mcg/kg/week — Peginterferon alpha-2b will be administered subcutaneously at a dose of 1.5 mcg/kg each week.
  Other Names: Pegintron®; Rebetol®
Drug: Ribavirin — Ribavirin will be administered orally at a dose of 800 mg/day to 1400 mg/day in two divided daily doses (BID).
  Other Names: Rebetol®; Pegintron®

SUMMARY:
This study is designed to assess the safety and tolerability of boceprevir dosed 800 mg three times daily (TID) orally (PO) in combination with Peginterferon alfa-2b (PEG2b) 1.5 mcg/kg once a week (QW) administered subcutaneously (SC) plus ribavirin (RBV) (800 to 1400 mg/day) PO in Response Guided Therapy (RGT) in adult Vietnamese subjects with Chronic Hepatitis C, Genotype 1 (CHC GT1) who failed prior treatment with any interferon and ribavirin in Vietnam.

DETAILED DESCRIPTION:
Each participant will participate in the trial for a maximum of 80 weeks from the time the participant signs the Informed Consent Form (ICF) through the final contact. After a Screening phase of approximately 4 to 8 weeks, each participant will receive treatment for approximately 36-48 weeks depending on response at Treatment Week 8.

A 4-week lead-in period with PEG2b plus RBV will be followed by 32 weeks boceprevir plus PEG2b/RBV. At treatment Week 36 participants will be assigned to the following treatments depending on the virologic response at Week 8 and cirrhotic status:

1. For non-cirrhotic participants with undetectable hepatitis C virus (HCV)-RNA on Week 8, all treatment will be discontinued at Week 36.
2. For non-cirrhotic participants with detectable HCV-RNA on Week 8, only boceprevir treatment will be discontinued at Week 36 and PEG2b and RBV treatment will continue to Week 48.
3. For cirrhotic participants, the boceprevir plus PEG2b/RBV treatment will continue to Week 48.

The study has a futility rule at Week 12 at which point all subjects with detectable HCV-RNA levels will be discontinued. All participants will have a post-treatment follow-up period of at least 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Weight ≥ 40 kg to ≤ 125 kg
* Sexually active male participants and female participants of child-bearing potential must agree to use a medically acceptable form of contraception
* Must have documented Chronic Hepatitis C Genotype 1 infection
* Must have failed prior treatment with interferon plus ribavirin
* Must have completed treatment with interferon plus ribavirin for at least 12 weeks
* Must have had a liver biopsy or Fibroscan to determine status as cirrhotic or non-cirrhotic
* Participants with cirrhosis must have had an ultrasound or imaging study within 6 months of the Screening visit

Exclusion Criteria:

* Known co-infection with the human immunodeficiency virus (HIV) or the hepatitis B virus
* Prior discontinuation of treatment with interferon or ribavirin due to the occurrence of an adverse event(s) considered by the investigator to be possibly or probably related to the treatment
* Treatment with ribavirin within 90 days and any interferon within 1 month of the Screening visit
* Treatment with any investigational drug within 30 days prior to the Screening visit
* Treatment with midazolam, pimozide, amiodarone, flecainide, propafenone, quinidine, or ergot derivatives within 2 weeks prior to the Day 1 visit
* Participation in any investigational trial within 30 days of the Screening visit
* Evidence of decompensated liver disease
* Child Pugh score > 6 (Class B and C)
* Diabetic and/or hypertensive participants with clinically significant ocular examination findings
* Pre-existing psychiatric conditions
* Clinical diagnosis of substance abuse
* Active or suspected malignancy
* Pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-05; Primary Completion 2016-09 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Achieving Sustained Virologic Response (SVR) | Follow-Up Week 24
Percentage of Participants Experiencing a Serious Adverse Event (SAE) During the Study Therapy Period | Treatment Week 1 to Treatment Week 24